CLINICAL TRIAL: NCT02418442
Title: Observational Study of Pediatric Rheumatic Diseases: The CARRA Registry
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Childhood Arthritis and Rheumatology Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00054616
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Rheumatic Joint Disease
Keywords: Systemic Arthritis; Oligoarthritis; Polyarthritis (Rheumatoid Factor Negative); Polyarthritis (Rheumatoid Factor Positive); Psoriatic Arthritis; Enthesitis Related Arthritis (ERA); Undifferianted Arthritis; CARRA Consensus Treatment Plans
MeSH Terms: conditions — Arthritis; Negative rheumatoid factor polyarthritis; Arthritis, Psoriatic; Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Biosample collection is active for a subset of subjects within the registry
Oversight: Data Monitoring Committee: No

SUMMARY:
Continuation of the CARRA Registry as described in the protocol will support data collection on patients with pediatric-onset rheumatic diseases. The CARRA Registry will form the basis for future CARRA studies. In particular, this observational registry will be used to answer pressing questions about therapeutics used to treat pediatric rheumatic diseases, including safety questions.

DETAILED DESCRIPTION:
The original Childhood Arthritis & Rheumatology Research Alliance (CARRA) Registry (Protocol Number: CRNT_REGST01) was first established in 2010 to advance alliance infrastructure, facilitate expanded clinical and translational pediatric research, and transform the culture of pediatric rheumatology toward universal participation in research. This original CARRA Registry will be referred to throughout the protocol as the CARRA Legacy Registry. Through the creation of a sophisticated informatics infrastructure, provision of comprehensive site support and the engagement of families, patients, and communities, the CARRA Registry will provide the opportunity for affected children at every CARRA Registry site to participate in high-quality clinical and translational research.

Continuation of the CARRA Registry as described in this protocol will support data collection on patients with pediatric-onset rheumatic diseases. The CARRA Registry will form the basis for future CARRA studies. In particular, this observational registry will be used to answer pressing questions about therapeutics used to treat pediatric rheumatic diseases, including examining safety questions. The Duke Clinical Research Institute (DCRI) is serving as the CARRA Clinical and Data Coordinating Center (CDCC) for the protocol.

Traditional exposure-based post-marketing registries of individual therapeutic agents for juvenile idiopathic arthritis (JIA), systemic lupus erythematosus, and other rheumatic diseases are inadequate for answering important safety questions for many reasons:

* Sample sizes are too small to detect uncommon but important events
* No unexposed comparators exist to evaluate risk attributable to underlying disease
* Duration of follow-up of individual patients is too short to evaluate many potential delayed adverse events (AEs)
* Sample sizes are inadequate to assess myriad complex and dynamic concurrent medication regimens common to treatment of rheumatic diseases
* Selective patient enrollment limits evaluation of co-morbid conditions and other patient factors

These limitations prevent patients, families, and providers from understanding the true risks and benefits of therapy in order to make appropriate and informed decisions. They also prevent drug manufacturers and regulatory agencies from conducting an informed review of marketed products for these diseases.

A registry based on disease diagnosis rather than specific therapeutic agents overcomes many of the limitations of exposure-based single-agent registries in the assessment of delayed or uncommon safety events. Indeed, data from a consolidated disease-based registry "...could provide the information necessary for individual companies to satisfy post-marketing requirements and commitments and obviate the need for an individual product registry" (letters from the United States (US) Food and Drug Administration (FDA) to CARRA, 21 December 2010 and 9 December 2011). This protocol details the foundation of a registry to meet these objectives.

The CARRA Registry aims to detect and understand the epidemiology of important AEs, including those that are delayed or uncommon. Subjects followed at active CARRA Registry sites are eligible for enrollment, regardless of past or current treatment. Each subject will be followed prospectively for a goal of 10 years duration; the study will continue indefinitely as resources allow and continued need exists. Data will be systematically collected, including important patient factors, therapies, serious adverse events (SAEs), and protocol-defined events of special interest. Selected safety events (e.g., malignancies) will be adjudicated by a panel of experts via a review of medical records. The CARRA Registry, a disease-based prospective observational registry, enables both detection of potential safety signals and hypothesis-driven, rigorous, and adequately-controlled pharmacoepidemiologic studies of important AEs and their associations with therapeutic agents.

In addition to answering questions about the safety of therapeutics, the data collected in the CARRA Registry are anticipated to serve many other valuable uses. Within the confines of observational study design, the effectiveness of therapeutic agents may be examined for short- and long-term clinical and patient-centered outcomes.

The Registry is the data collection platform for Consensus Treatment Plan (CTP) comparative effectiveness research in pediatric rheumatic disease. Patients enrolled in the Registry may also be eligible to be followed as part of a CTP subset. Examples of CTP projects include:

FiRst line Options for Systemic JIA Treatment (FROST). The purpose of FROST was to compare the effectiveness of CARRA systemic JIA (sJIA) treatment strategies (biologic vs. non-biologic) in achieving clinically inactive disease in patients with new-onset sJIA. Additionally, FROST aimed to compare patient/caregiver reported outcomes between treatment strategies. FROST enrolled new-onset, previously untreated sJIA patients who are starting treatment with one of the 4 sJIA CTPs (glucocorticoid (GC) only; Methotrexate + GC; IL-1 inhibitor + GC; IL-6 + GC). Enrollment will occur over 3 years at all CARRA Registry sites. In addition to routine Registry data collection, patients followed as part of the FROST CTP completed additional questionnaires about their disease status and quality of life.

Medication use for pediatric rheumatic diseases is dynamic and not well characterized. The CARRA Registry represents a powerful data source to follow drug use patterns and provides the opportunity to study predictors of medication use. Important outcomes are likely to be influenced by other factors in addition to therapy (e.g., disease severity) and the CARRA Registry is positioned to help answer these types of questions. Patient-reported outcomes (PROs) generated by patients outside the context of clinical encounters may be collected in the Registry to provide a rich, additional dimension of data to better understand rheumatic diseases. Practitioners may review clinical data from their sites as part of a quality improvement approach to better outcomes.

Analyses of CARRA Registry data aim to provide results to guide the therapeutic decisions made by affected children, families, and providers while improving regulatory efficiency and reducing cost. Ultimately, this approach might serve as a model for successful collaboration between research community networks, industry, and public agencies to promote the effective and efficient evaluation of drugs and devices across the regulatory continuum.

ELIGIBILITY:
Inclusion Criteria:

1. Onset of rheumatic disease prior to age 16 years for JIA and onset prior to age 19 years for all other rheumatic diseases (see appendix A).
2. Subject (and/or parent/legal guardian when required) is able to provide written informed consent and willing to comply with study procedures.
3. Subject and/or parent/legal guardian is willing to be contacted in the future by study staff.

Exclusion Criteria:

1. Greater than 21 years of age at the time of enrollment.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with pediatric rheumatic diseases enrolled from participating CARRA sites.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2015-07; Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Prospectively collect essential data elements from children, adolescents and young adults with pediatric rheumatic diseases | Approximately 10 years
Evaluate the safety of therapeutic agents in persons with pediatric onset rheumatic diseases | Approximately 10 years

SECONDARY OUTCOMES:
Evaluate clinical outcomes associated with the use of therapeutic agents in persons with pediatric onset rheumatic diseases | Approximately 10 years
Document drug treatment patterns and clinical course of persons with pediatric onset rheumatic diseases over time. | Approximately 10 years
Evaluate factors other than drug treatments that are associated with clinical outcomes in pediatric onset rheumatic diseases | Approximately 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Mara L Becker, MD, MSCE, Principal Investigator — Duke Clinical Research Insitute; Mary Beth Son, MD, Principal Investigator — Boston Children's Hospital; Timothy Beukelman, MD, MSCE, Principal Investigator — University of Alabama at Birmingham
Locations (82):
- United States (75):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Mattel Children's Hospital at University of California Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital San Diego, San Diego, California
  - University of California at San Francisco Medical Center, San Francisco, California
  - The Children's Hospital of Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - University of Florida - Shand's Children's Hospital, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Georgia Regents University Medical Center, Augusta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - The University of Iowa Hospitals and Clinics (University of Iowa Children's Hospital), Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville Schoole of Medicine, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital for Children, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Bay State Medical Center, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Helen Devos Children's Hospital, Grand Rapids, Michigan
  - West Michigan Rheumatology, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Saint Louis University School of Medicine, St Louis, Missouri
  - Saint Louis Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Goryeb Children's Hospital, Morristown, New Jersey
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - The Pediatric Specialty Center at Saint Barnabas, West Orange, New Jersey
  - Albany Medical College, Albany, New York
  - Cohen Children's Medical Center of New York, Lake Success, New York
  - New York University Langone Medical Center, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - Children's Hospital at Montefiore, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Levine Children's Hospital / Carolinas Medical Center, Charlotte, North Carolina
  - Duke Children's Hospital & Health Center, Durham, North Carolina
  - Wake Forest Baptist Brenner Children's Hospital, Winston-Salem, North Carolina
  - Sanford Health, Fargo, North Dakota
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - UH Rainbox Babies and Children's Hospital, Cleveland, Ohio
  - Metrohealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Randall Children's Hospital at Legacy Emanuel, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh UPMC, Pittsburgh, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Medical University of South Carolina Children's Hospital, Charleston, South Carolina
  - Monroe Carrell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - University of Texas Southwestern Medical Center Dallas, Dallas, Texas
  - Baylor College of Medicine Pediatric Immunology Allergy Rheumatology, Houston, Texas
  - University of Utah Hospitals and Clinics (Primary Children's Hospital), Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin, American Family Children's Hospital, Madison, Wisconsin
  - Children's Hospital Of Wisconsin, Wauwatosa, Wisconsin
- Canada (4):
  - University of Calgary - Alberta Children's Hospital, Calgary, Alberta
  - University of Manitoba - Children's Hospital of Manitoba, Winnipeg, Manitoba
  - IWK Health Center, Halifax, Nova Scotia
  - The Hospital for Sick Children, Toronto, Ontario
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel
- IRCCS Ospedale Pediatrico Bambino Gesu (OPBG), Rome, Italy
- San Jorge Children's Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Nigrovic PA, Beukelman T, Tomlinson G, Feldman BM, Schanberg LE, Kimura Y; Childhood Arthritis and Rheumatology Research Alliance Systemic Juvenile Idiopathic Arthritis Consensus Treatment Plan Workgroup. Bayesian comparative effectiveness study of four consensus treatment plans for initial management of systemic juvenile idiopathic arthritis: FiRst-Line Options for Systemic juvenile idiopathic arthritis Treatment (FROST). Clin Trials. 2018 Jun;15(3):268-277. doi: 10.1177/1740774518761367. Epub 2018 Mar 15. PMID 29542334